CLINICAL TRIAL: NCT01814943
Title: The Risk of Uncomplicated Peptic Ulcer in a Cohort of Secondary Prevention Aspirin Users
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5040N00007
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Uncomplicated Peptic Ulcer
Keywords: Uncomplicated peptic ulcer; Acid-suppressing drugs; Epidemiology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with prescription for low dose ASA (75-300 mg/day)

SUMMARY:
This study is conducted in a cohort of low dose aspirin (ASA) users previously ascertained. The aims of the post hoc analyses are:

To estimate the incidence of uncomplicated peptic ulcer (UPU) in a cohort of low-dose ASA for secondary prevention of vascular disease and the relative risk of UPU associated with use and discontinuation of use of low dose ASA.

To estimate the effect of proton pump inhibitors (PPI) on the occurrence of UPU among users of low-dose ASA for secondary prevention of vascular disease To evaluate the effect of other risk factors on the occurrence of UPU among users of low-dose ASA for secondary prevention of vascular disease.

DETAILED DESCRIPTION:
The risk of uncomplicated peptic ulcer in a cohort of secondary prevention aspirin users

ELIGIBILITY:
Inclusion Criteria:

- Patients aged 50-84 years in 2000-2007 with a first prescription of low dose ASA ( see study population description)

Exclusion Criteria:

- Patients aged below age 50 and 85 years and above ( see study population description)

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 50-84 yrs who had a first prescription of low-dose ASA (75-300mg/day) for secondary cardiovascular or cerebrovascular prevention in 2000-2007 in The Health Improvement Network database in the UK. Patients had to be enrolled with their PCP (Primary Care Physician) for at least 2 years and have a health contact in the year prior. Patients with use of aspirin ever recorded in the database before start of follow-up as well as patient with cancer or alcohol abuse were excluded. Individuals were followed up until the earliest occurrence of one of the following endpoints; first recorded diagnosis of uncomplicated peptic ulcer, canser, alcohol abuse or alcohol related disease, reaching the age of 85 years old, date of last practice data collection, death or end of follow-up ( 30 September 2011).Patient records were manually reviewed to validate cases.
Sampling Method: Non-Probability Sample
Enrollment: 39000 (Actual)
Dates: Start 2012-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incidence rates of uncomplicated peptic ulcer in a cohort of secondary prevention aspirin users | From 1 January 2000 till 30 September 2011, an expected average of 6 years.
Risk (hazard ratio) of developing uncomplicated peptic ulcer in a cohort of secondary prevention aspirin users | From 1 Januart 2000 till 30 September 2011, an expected average of 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Garcia Rodriguez, MD, Principal Investigator — CEIFE (Centro Espanol de Investigacion Farmacoepidemiologica - Spanish Centre for Pharmacoepidemiologic Research )
Locations (1):
- Research Site, Madrid, Spain

REFERENCES:
- [Background] Cea Soriano L, Rodriguez LA. Risk of Upper Gastrointestinal Bleeding in a Cohort of New Users of Low-Dose ASA for Secondary Prevention of Cardiovascular Outcomes. Front Pharmacol. 2010 Oct 14;1:126. doi: 10.3389/fphar.2010.00126. eCollection 2010. PMID 21811460
- [Background] Garcia Rodriguez LA, Cea Soriano L, Hill C, Johansson S. Increased risk of stroke after discontinuation of acetylsalicylic acid: a UK primary care study. Neurology. 2011 Feb 22;76(8):740-6. doi: 10.1212/WNL.0b013e31820d62b5. Epub 2011 Jan 26. PMID 21270415